CLINICAL TRIAL: NCT05022693
Title: An Open-Label, Single-Dose Pharmacokinetic Study of Liquid Subcutaneous Formulation of BIO89-100 in Subjects With Nonalcoholic Steatohepatitis (NASH) With Compensated Cirrhosis
Brief Title: PK Study of Liquid Formulation of BIO89-100 in Subjects With NASH With Compensation Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 89bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BIO89-100-111
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Open label, single dose, PK study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BIO89-100 30 mg, Open Lable, Single Dose (Experimental)
  Interventions: Drug: BIO89-100

INTERVENTIONS:
Drug: BIO89-100 — Subcutaneous Injections

SUMMARY:
This is an open-label, single-dose study to evaluate the PK profile of the liquid SC formulation of BIO89-100 in approximately 8 male and female subjects with NASH with compensated cirrhosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 21 to 65
* Diagnosis of NASH with compensated cirrhosis by a hepatologist based on Liver Forum criteria.
* Model for End-Stage Liver Disease (MELD) score < 12.
* Child-Turcotte-Pugh (CTP) score < 7 (Class A).
* Fibrosis stage F4 by FibroScan.

Key Exclusion Criteria:

* History of hepatic cirrhosis decompensation, OR overt hepatic encephalopathy OR signs of hepatic cirrhosis decompensation.
* Prior transjugular intrahepatic portosystemic (TIPS) shunt procedure.
* known condition other than cirrhosis that may possibly interfere with drug absorption, distribution, metabolism, or excretion.
* Significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
PK Profile of liquid formulation of BIO89-100 | 22 days
  Determine maximum observed serum drug concentration (Cmax)
PK Profile of liquid formulation of BIO89-100 | 22 days
  Area under the serum drug concentration-by-time curve from time 0 to the time of the last quantifiable drug concentration (AUC0-t)

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of the BIO89-100 liquid formulation | 22 days
  Frequency and severity of adverse events (AEs) and serious adverse events (SAEs)
  Number of subjects who discontinued due to AEs and due to related AEs

CONTACTS AND LOCATIONS:
Locations (1):
- 89bio Clinical Study Site, Chandler, Arizona, United States